CLINICAL TRIAL: NCT03179826
Title: Analysis of Inhaled Corticoid Prescriptions in General Medicine
Acronym: COMEGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17-0152; 2017-A01230-53 (Other: RCB number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Adults consulting with one of the participating general practitioners and requiring long term inhaled corticoids and monitoring.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and asthma are frequent and disabling pathologies. The general practitioner is often at the front line vis-a-vis screening, diagnosis and treatment of these pathologies. There are currently many treatments available, in particular inhaled corticosteroids, and although the recommendations for management appear to be well codified in theory, the adaptation of drug therapy remains complex in general practice.

The prescription of inhaled corticosteroids, often initiated during a general medicine consultation, is not simple. The aim of this study is to analyze the relevance of the prescription of inhaled corticosteroids in primary care and to identify the criteria necessary for the prescription of inhaled corticosteroids available in general practice.

The main objective of our study is to evaluate the rate of consultations where all the elements required for guiding the prescription of an inhaled corticoid are available.

The secondary objectives are:

* Identify other factors associated with decision-making
* Identify the causes of inhaled corticosteroid stopping (de-prescription)

ELIGIBILITY:
Inclusion Criteria:

* Patient with short-term inhaled corticosteroid therapy
* Informed and not opposed to participate in this research

Exclusion Criteria:

* Patient under judicial or legal protection
* Adults under any kind of guardianship -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adults consulting with one of the participating general practitioners and requiring long term inhaled corticoids and monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of all factors justifying the prescription of inhaled cortcoids | Day 0 (transversal study)
  The presence (yes/no) of all factors justifying the prescription of inhaled cortcoids as described in the associated market authorization.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — Montpellier University Hospitals
Locations (2):
- France (2):
  - Cabinet de médecine générale, Clapiers
  - Cabinet de médecine générale, Saint-Martin-de-Londres